CLINICAL TRIAL: NCT06668428
Title: Effects of Virtual Reality and Nature Sounds on Pain and Anxiety After Cesarean Section: A Randomized Controlled Trial
Brief Title: Effects of Virtual Reality and Nature Sounds on Pain and Anxiety in Women Having Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nazlı Baltacı, Associate Professor, phD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMU-TURKMEN-2024/367
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Obstetrics and Gynaecology; Nursing; Caesarean Section; Pain; Anxiety
Keywords: Pain; Anxiety; Caesarean Section; Nurse; Virtual Reality; Nature Sounds
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a two-group, parallel, randomized, controlled experimental study with a pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group with Standard Care (No Intervention): Participants in the control group did not undergo any intervention other than routine post-caesarean care (verbal information about the procedure and brief written information about the procedure are planned to be provided).
- Control Group Using Virtual Reality Glasses (Experimental): The researcher informed the women in the intervention group about the study, introduced them to the virtual reality glasses after obtaining written consent, and taught them how to use the glasses. Subsequently, the data collection form, State Anxiety Scale, and visual analogue scale rating scale for pain were administered face-to-face to both groups. After the first mobilisation, postpartum women were shown a nature landscape video through virtual reality glasses (VRG) accompanied by nature sounds for an average of 20 minutes. Each woman watched the same video. Pain and anxiety were reassessed after the application. The same application was performed for each woman, and the goggles were disinfected with Dermosept surface disinfectant, which provides cold sterilisation, prior to the application.
  Interventions: Device: Virtual Reality Glasses

INTERVENTIONS:
Device: Virtual Reality Glasses — Pharmacological and non-pharmacological methods are applied in the management of pain and anxiety after cesarean section (Tetik & Tekinemre, 2017). In addition to medical treatment during the post-cesarean care process, complementary and supportive non-pharmacological approaches can be used to address the woman holistically and provide multi-faceted contributions to the health of the mother and baby (Ali, 2022; Bayraktar, 2023). One of the non-pharmacological approaches, virtual reality glasses, is a device that provides two or three-dimensional environments to stimulate our senses by creating illusions of images (Appel et al., 2021). SGG creates a therapeutic effect by diverting attention, provides relaxation, and can thus be used in the management of pain and anxiety (Ayed et al., 2019). It has been determined that virtual reality glasses are an effective method in the management of pain and anxiety in the field of nursing (Akıncı & Aydın Özkan, 2024).
  Arms: Control Group Using Virtual Reality Glasses

SUMMARY:
This study was conducted to determine the effects of virtual reality application on pain and anxiety in women who gave birth by caesarean section. It was applied to women who had given birth by caesarean section at a public hospital in northern Turkey, voluntarily agreed to participate in the study, and were randomly assigned to the intervention (n=40) and control (n=40) groups. Women in the intervention group were taught how to use virtual reality goggles. After the first mobilisation, women were shown a nature landscape video through virtual reality goggles (VRG) accompanied by nature sounds for an average of 20 minutes. The aim of this application was to enable women to view nature images more effectively accompanied by nature sounds, thereby helping them to focus on the images and sounds, distract their attention, relax, and escape the tension of their surroundings. The application was carried out with the women in a semi-reclining position and without sleeping. The same application was applied to each woman, and the glasses were disinfected with Dermosept surface disinfectant, which provides cold sterilisation, before the application. No application was made to the women in the control group; only the hospital's routine care was applied. The data were collected by the researcher through face-to-face interviews based on the statements of women after caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being over 18 years of ageBeing able to read and write in Turkish
* Giving birth at term, having a single, live and healthy baby
* The baby being with the mother
* Having a healthy/risk-free pregnancy
* Having had spinal anesthesia.

Exclusion Criteria:

* Having a diagnosed psychiatric disease,
* Having a mental disability and communication problem,
* Having a vision or hearing problem,
* Developing complications during or after a cesarean section,
* Having any obstacles to postpartum mobilization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 80 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
State Anxiety Level | Anxiety levels were assessed before and after the intervention.
  State anxiety level will be measured with Spielberger State Anxiety Scale. The Turkish reliability and validity study of the scale, which was developed by Spielberger and his colleagues to measure an individual's state and trait anxiety levels, was conducted by Öner and Le Compte in 1983. The scale examines anxiety in two sub-dimensions: State Anxiety measures an individual's feelings under a certain moment and condition, while Trait Anxiety expresses the individual's general anxiety level. Each statement in the scale is a 4-point Likert-type scale. There are 20 items in both types in the Spielberger State-Trait Anxiety Scale. The total score obtained from the scale varies between 20 and 80, with high scores indicating a high level of anxiety. The scale does not have any cut-off value. Cronbach's alpha coefficient was found to be 0.83 for State Anxiety.
Pain Level | Pain levels were assessed before and after the intervention.
  Pain level will be measured with Visual Analog Scale. The use of the scale, developed by Price et al. in 1983, is achieved by measuring pain based on the statements of the people participating in the research. It is a one-dimensional, easy-to-administer scale and is widely used. It is a scale that the individual evaluates by making marks on a horizontal or vertical line of 10 cm or 100 mm, indicating that one end is very good and the other end is very poor. In our study, the scale starts with "mild pain" and ends with "very severe pain". A higher score from the scale indicates increased pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Baltacı, Assoc. Prof., phD, Study Director — baltacinazli@gmail.com; Gizem Türkmen, MSc Student, Principal Investigator — gizemturkkmen19@gmail.com
Locations (1):
- Gynecology and Obstetrics Department affiliated to the Gynecology and Obstetrics Department of Samsun Education and Research Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
You are undertaking that your answers to the questions will be kept confidential and will not be shared with anyone.